CLINICAL TRIAL: NCT07007468
Title: The Effect of Abdominal Massage in Prevention of Chemotherapy-Induced Constipation
Brief Title: Prevention of Constipation in Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: İUC-FNHF-CL-01
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Constipation Drug Induced
Keywords: chemotherapy; constipation; massage
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: two groups with a conventional therapy control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Massage Group (Experimental): Patients will be informed about the abdominal massage application; they will be informed that it should be applied twice a day for five days, 30 minutes after breakfast for 15 minutes and 30 minutes after dinner for 15 minutes. In order to make the massage application more understandable and effective, the abdominal massage application video to be created by the researcher will be shared with the patient and his/her family. After the fifth day of the Abdominal Massage application, patients will be evaluated for the last time with the Bristol Stool Consistency Scale (Appendix-2), Constipation Severity Scale (Appendix-3), Constipation Quality of Life Scale (Appendix-4) and Patient Monitoring and Control Form (Appendix-5).
  Interventions: Other: Abdominal Massage
- Control Group (No Intervention): Patients who were determined to have constipation as a result of the Bristol Stool Consistency Scale evaluation and assigned to the control group by randomization method will first be administered the Patient Identification Form (Appendix-1), Constipation Severity Scale (Appendix-3), Constipation Quality of Life Scale (Appendix-4), and Patient Monitoring and Control Form (Appendix-5). The researcher will provide information about the "Patient Follow-up and Control Form (Appendix-5)" and the patients will be followed up regularly for five days.
  After five days of follow-up, the patients will be evaluated with the Bristol Stool Consistency Scale (Appendix-2), Constipation Severity Scale (Appendix-3), Constipation Quality of Life Scale (Appendix-4) and Patient Follow-up and Control Form (Appendix-5).

INTERVENTIONS:
Other: Abdominal Massage — Abdominal massage is a massage technique performed with soft and rhythmic movements applied to the abdomen. Abdominal massage is an inexpensive, non-invasive, non-harmful, non-invasive method that can be applied by nurses for the treatment of constipation or by teaching the patient and his/her family. During the application of abdominal massage, effleurage (patting), abdominal effleurage , petrissage (kneading), abdominal petrissage maneuvers are applied.
  Arms: Abdominal Massage Group

SUMMARY:
Constipation is the third most common symptom in patients undergoing chemotherapy, with an incidence rate ranging from 31% to 90%. Despite its high prevalence and adverse effects on patients, constipation is often not reported by patients and is not frequently monitored by nurses, resulting in delays in treatment and care. Prolonged constipation can lead to health problems such as fecal impaction/obstruction, hemorrhoids, rectal pain, and intestinal perforation, thereby reducing patients' quality of life. Additionally, increased severity of constipation in cancer patients may lead to the interruption or complete cessation of chemotherapy. Therefore, it is essential to monitor and assess patients for the risk of developing constipation and to implement an effective nursing care protocol.

Abdominal massage is an approach that increases peristalsis, i.e., digestive system movement, by altering intra-abdominal pressure, thereby reducing the severity of constipation.

DETAILED DESCRIPTION:
Cancer is one of the most important health problems in our country and in the world. According to the Global Cancer Observation Data (GLOBOCAN), 9.7 million people lost their lives due to cancer in 2022. There are many methods such as chemotherapy, radiotherapy and surgical treatment in the treatment of cancer. Chemotherapy is the most commonly used of these systemic treatment approaches. Chemotherapy-related gastrointestinal symptoms such as constipation, diarrhea, bloating, incontinence, flatulence and abdominal distension are observed in patients. Constipation is the third most symptom in patients receiving chemotherapy, with a prevalence of 40% to 90%.

Although constipation is common and affects patients negatively, it is not expressed by patients and is not frequently followed up by nurses, resulting in disruptions in the treatment and care process. Prolongation of the constipation process health problems such as fecal impaction / obstruction, hemorrhoids, rectal pain and intestinal perforation and decreases the quality of life of the patients. In addition, increased severity of constipation in cancer patients leads to interruption or complete termination of chemotherapy. Therefore, patients be monitored and evaluated in terms of the risk of constipation development and an effective nursing care protocol should be implemented.

Pharmacologic, non-pharmacologic and surgical methods are used to prevent constipation. Pharmacologic and surgical approaches are quite costly. In the non-pharmacological approach; methods such as increasing fiber food and water consumption, regular exercise, abdominal massage are used. Abdominal massage is a non-invasive nonpharmacologic approach that increases digestive system movement by changing intra-abdominal pressure, reduces the severity of constipation, is safe and has no side effects, and can be applied by nurses with independent decision-making authority and educator role.

This thesis was planned to evaluate "The Effect of Abdominal Massage in the Prevention of Chemotherapy Associated Constipation".

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Receiving chemotherapy for breast cancer or lung cancer that causes constipation
* Patients who received at least one cycle of chemotherapy and experienced chemotherapy-associated constipation within five days of treatment (stool type 1 or 2 according to the Bristol Stool Scale)
* Volunteers who are willing to participate in the research, can communicate, and can read and write,
* Without psychiatric illness and abdominal obstruction,
* No mass in the abdominal region was detected,
* No intestinal bleeding,
* No history of radiation therapy to the abdominal region,
* No surgical procedures in the abdominal region,
* Patients without intra-abdominal infection, inflammatory bowel disease and irritable bowel syndrome will be included

Exclusion Criteria:

* Patients with stool type 3, 4, 5, 6 and 7 points according to the Bristol Stool Scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Identification Form | one day
  This form was created by the researcher by reviewing the literature. The form included a total of 39 questions about the patient's current disease, descriptive characteristics, socio-demographic characteristics, chemotherapy cycle and regimen, medication use that may cause constipation, performance status score, appetite status, amount of fluid consumed daily, physical activity status, and food group consumed in the last week.
Bristol Fecal Consistency Scale | five days
  The Bristol Stool Consistency Scale was developed by Lewis et al. The form of the stool varies according to the transit time through the intestine. With this scale, the stool form is evaluated over seven different stool types. In the scale, 1 and 2 points are evaluated as "hard stool-constipation", 3, 4 and 5 points as "normal stool", 6 and 7 points as "soft-watery stool (diarrhea)".
Constipation Severity Scale | two days
  The Constipation Severity Scale (CSS) was developed by Varma et al. in 2008. Its Turkish validity and reliability was performed by Kaya. The scale consists of 16 items to determine the frequency and intensity of defecation and difficulty/difficulty during defecation. The scale has 3 sub-dimensions: "fecal obstruction", "laziness of the large intestine" and "pain". The score that can be obtained from the fecal obstruction sub-dimension is between 0-28, the score that can be obtained from the large intestine sub-dimension is between 0-29, and the score that can be obtained from the pain sub-dimension is between 0-16. The lowest total score that can be obtained from the scale is 0 and the highest score is 73. A high score on the scale indicates that the symptoms are serious. Cronbach's alpha value of the original scale: 0.88-0.91; Cronbach's alpha of the Turkish scale: 0.92-0.93.
Constipation Quality of Life Scale | two days
  The scale, which was developed by Marquis et al. (2005), and validated and reliably analyzed in Turkish (2015), consists of a total of 28 items. This five-point Likert scale consists of 4 sections: 'Anxiety or Worry' (11 items), 'Physical Discomfort' (4 items), 'Psychosocial Discomfort' (8 items) and 'Satisfaction' (5 items). In the Constipation Quality of Life Scale, questions 18, 25, 26, 27 and 28 are reverse items and are calculated by reversing them. A minimum score of 28 and a maximum score of 140 is obtained from this scale. The Cronbach's alpha value of the scale is 0.96. A low total score indicates a high quality of life.
Patient Monitoring and Control Form | five days
  It is a simple, easy-to-implement, practical form created by the researcher to monitor the daily nutrients consumed by the patients, to monitor whether abdominal massage is performed, and to ensure that the Bristol Stool Consistency Scale (Appendix-2) evaluations are followed up by the patients and their families.

CONTACTS AND LOCATIONS:
Overall Officials: Can LAFÇI, PhD(c), Study Director — İSTANBUL
Locations (1):
- Istanbul University-Cerrahpasa Florence Nightingale Faculty of Nursing, Istanbul, Marmara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No